CLINICAL TRIAL: NCT05772910
Title: Viability of an Educational Program for Lifestyle Changes and an Algorithm for the Derivation of Exercise Programs in Older People at Risk of Dependency at Primary Care.
Acronym: PRICA-POWFRAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Alejandro Galán Mercant, Associate Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR2022-018
Record Dates: First submitted 2023-02-22; First posted 2023-03-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Frailty; Disability Physical; Old Age; Atrophy
Keywords: Education; Physical Exercise; Aging; Frailty; Dependency; Biomarkers; Older Adults; Machine Learning
MeSH Terms: conditions — Frailty; Atrophy; Motor Activity | interventions — Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EDUcation (Experimental): The EDU group will assist to an individualized educative program based on intrinsic capacity optimization through lifestyle changes.
  Interventions: Behavioral: EDUcation
- EXERcise (Experimental): The EXER group will follow a program focused on the specific deficit of muscular power from a simple clinical test such as the STS and, in addition, they will be evaluated to be able to prescribe training individually (evaluation of training)
  Interventions: Other: EXERcise
- EDU-EXER (Experimental): EDU-EXER group subject develops both interventions together.
  Interventions: Other: EDU-EXER
- CONtrol (Active Comparator): CON group will continue the usual clinical treatment and their normal life.
  Interventions: Other: CONtrol

INTERVENTIONS:
Behavioral: EDUcation — The education intervention will consist of an individualized educative program based on intrinsic capacity optimization through lifestyle changes. To develop the program, the program creation team will be multidisciplinary (psychologists, medical doctor, dietitian…) and will discuss goal setting, the education strategy, and retention of motivation. The experts are required to create the education program such that the participants can manage their health by themselves. The goal will be self-management of dietary habits and increases in physical activity levels for each individual case. The education program will be in Spanish or in English; as it will consist in personal counselling, even with a low level of the language the communication will be possible. The nutritional education program will be conducted every 2 weeks for 10 consecutive weeks, with 20-min counselling sessions by an expert.
  Other Names: EDU
  Arms: EDUcation
Other: EXERcise — The intervention period will have 10 weeks, in which the EXER group will carry out 2-3 sessions a week (total of 20-30 sessions). In this concurrent program, exercises of the lower extremities (leg press, abduction and plantar flexion) will be performed mainly on weight training machines. Intensity in each exercise will be individualized for each participant through a test to determine muscle power. In addition, in the last part of each session the participants will perform an endurance training type high insensitive interval training on a cycle ergometer (60-80 rpm). The intensity will be individualized to each patient through an incremental stress test until volitional exhaustion, and the subjects will alternate intervals of 30 seconds at 90% of the maximum workload, with intervals of 90 seconds at 40% of the maximum. Each session is estimated to have a total duration of 30-50 minutes.
  Other Names: EXER
  Arms: EXERcise
Other: EDU-EXER — This group will carry out the same two previous interventions together.
  Arms: EDU-EXER
Other: CONtrol — CONtrol group will continue the usual clinical treatment and their normal life
  Arms: CONtrol

SUMMARY:
According to the INE in 2021, more than 9 million people are currently over 65 years of age. This means that more than 1 million are frail and almost 4 million are pre-fragile only in Spain. Frailty is the prelude to disability and dependency, but unlike these, it is treatable and preventable. Currently, it is known that the best treatment for frailty is physical exercise and physical activity. The problem arises from the need that exists in the health system to prescribe individualized and patient-centered exercise, with the use of scarce resources (time, personnel, tools) and in a simple way in clinical practice. Additionally, the system needs tools that help us know (and predict) if this exercise prescription is efficient. Furthermore, frailty is a multidimensional syndrome, for which a comprehensive approach is necessary. The combined study of blood and digital biomarkers, as well as the plethora of dimensions evaluated (muscle and physical activity, cognitive, lifestyle, clinical, body composition, social, sleep), constitute an optimal approach that would provide a unique opportunity to understand prevention and treatment of unsuccessful aging and frailty. The PRICA-POWFRAIL project aims to examine the feasibility of an educational intervention to change lifestyle habits as well as the effect of a referral algorithm to an exercise program and lifestyle changes focused on treating specific deficits of low muscle power, powerful predictor of adverse health events. The subsequent referral will be implemented in a supervised exercise program at the functional, cognitive muscle level and in older people at risk of dependence. Secondarily, the effect of this intervention on blood biomarkers (at a genetic, epigenetic and metabolomic level), physical health (functional capacity, blood pressure, body composition) and mental health (quality of life and depression), as well as on other risk factors (genetic and biological) for the development of frailty. A total of 110 people older than 70 years of age in previous stages of dependency will be randomly distributed among the group of an educational program, the intervention group with supervised physical exercise, a intervention group with both previous educational and exercise programs and the control group. The design will include a 10- week intervention with pre and post-intervention measurement phases and a third measurement (retest) 12 months after completion. The supervised physical exercise program will be of a multi-component type including cardiovascular, muscular, coordinative and balance work, and a progression will be established in the different load parameters (frequency, volume, intensity, density). This will allow us to understand from a very complete perspective the causes and mechanisms underlying this response. The PRICA-POWFRAIL project Will mean a significant increase in scientific knowledge about the response and response rate to ultra-individualized exercise programs directed as a therapeutic measure in people at risk of dependency from a multidimensional perspective. In addition, the project will have a relevant impact at the social and economic level by transferring the findings of the study to the social and health field through the agents and means provided in it.

ELIGIBILITY:
Inclusion Criteria:

Following the 2014 Consensus Document on the prevention of frailty and falls in the elderly patient we will recruit individuals

I) > 70 years of age

II) with a Barthel Index score > 75

III) meeting at least one of the following two criteria: a score ≤9 in the short physical performance battery (SPPB) or FRAIL questionnaire with values 1 or 2.

Exclusion Criteria:

I) Inability to go to the Primary Care Health Centre for any reason.

II) Moderate to severe cognitive impairment (Mini-Mental State Examination< 20 points

III) Severe pathology for which physical activity is contraindicated at the physician's discretion including but not limited to: recent acute myocardial infarction (6 months), uncontrolled cardiac arrhythmia, severe cardiac valve disease, non-controlled hypertension (> 180/100mmHg), non-controlled/severe heart failure, severe respiratory insufficiency disease, and diabetes mellitus with acute decompensation/frequent hypoglycaemia.

Ages: 70 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Relative lower limbs muscle power | Change from Baseline STS muscle power at 12 weeks
  The STS muscle power test was used to assess mechanical power. Participants were instructed to perform 5 timed STS repetitions after the cue "ready, set, go!", as fast as possible, on a standardized armless chair (height = 0.43 m) with arms crossed over the chest. Importantly, from the sitting position, they had to fully extend their knees and hips to the standing position, and descend to the sitting position until at least touching the chair with their buttocks. The test was repeated when any of these instructions was broken. The time (±0.01 s) needed to perform 5 STS repetitions was recorded using a stopwatch. Absolute STS muscle power (W) was calculated using an equation where body mass is indicated in kg, body height and chair height in m, and five STS time in s (Alcazar et al. 2018).
  Alcazar, J. et al. The sit-to-stand muscle power test: An easy, inexpensive and portable procedure to assess muscle power in older people. Exp Gerontol 112, 38-43 (2018).
Vital functional capacity | Change from Baseline Vital functional capacity at 12 weeks
  The vital functional capacity will be evaluated through cardiorespiratory function using an indirect test adapted to the age range (field tests, which allow obtaining an estimated value of maximum oxygen consumption, the best integral marker of the physiological reserve of an individual, namely 6minute walking test or the 2 min-version which is highly correlated.
Level of physical activity during the daily life | Change from Baseline Level of physical activity at 12 weeks
  Measured by accelerometry for 1 week in evaluation timepoints.

SECONDARY OUTCOMES:
The quality of life (QoL) | Change from Baseline the quality of life at 12 weeks
  EQ-5D which measures health-related QoL through physical, psychological and social dimensions.
Subjective health-status level | Change from Baseline the health status level at 12 weeks
  SF-36 questionnaire which measures the subjective health-status level.
Cognitive Function - Mini-mental state examination (MMSE) | Change from Baseline MMSE at 12 weeks
  The mini-mental test is a simple test that allows detecting the presence of cognitive impairment, that is, of dementia. It can be normal in people with mild cognitive impairment or with incipient forms of Alzheimer's requiring, in these cases, studies with more sophisticated tests.
Cognitive Function - The Montreal cognitive assessment test (MoCA) | Change from Baseline MoCA at 12 weeks
  The Montreal cognitive assessment test (MoCA) is a brief instrument with which, in a specific way, mild cognitive impairment is detected, as well as dementia.
Mood State - Geriatric Depression Scale (GDS) | Change from Baseline Geriatric Depression Scale (GDS) at 12 weeks
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. The GDS was originally developed as a 30-item instrument. Since this version proved both time-consuming and difficult for some patients to complete, a 15-item version was developed.
Nutritional profile measurements - Mediterranean Diet Adherence Screener index | Change from Baseline Nutritional profile at 12 weeks
  1. MEDAS (Mediterranean Diet Adherence Screener index). Scale of adherence to the Mediterranean diet of 14 items.
Degree of frailty - Fried criteria | Change from Baseline frailty degree at 12 weeks
  The Fried frailty phenotype (FP) assesses physical frailty through five criteria: unintentional weight loss; weakness or poor handgrip strength; self-reported exhaustion; slow walking speed; and low physical activity.
Body composition - Bioimpedance | Change from Baseline Bioimpedance composition at 12 weeks
  The body composition will be evaluated by means of bioimpedance.
Body composition - body mass index (BMI) | Change from Baseline body mass index (BMI) at 12 weeks
  Weight and height will be combined to report BMI in kg/m^2
Body composition - height | Change from Baseline height at 12 weeks
  Height measure in meter
Body composition - weight | Change from Baseline weight at 12 weeks
  Weight measure in kilograms
Musculoskeletal ultrasound architecture | Change from Baseline Musculoskeletal ultrasound architecture at 12 weeks
  All ultrasound images will be acquired by the same operator with the same ultrasound device throughout the whole study using a linear 40 mm transducer and a phased array transductor, and images will be analysed through the ACSAuto script to semi-automatically evaluate ultrasound pictures. The vastus lateralis architecture will be analysed through the Simple Muscle Architecture Analysis tool for Fiji. These procedures will be done according to Rodriguez-López et al.
  Rodriguez-Lopez, C. et al. Effects of Power-Oriented Resistance Training With Heavy vs. Light Loads on Muscle-Tendon Function in Older Adults: A Study Protocol for a Randomized Controlled Trial. Front Physiol 12, (2021).
Depressive Symptoms | Change from Baseline Depressive Symptoms at 12 weeks
  The depressive symptoms will be assessed with the Geriatric Depression scale to assess psychology status of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Galan-Mercant, PhD, Principal Investigator — University of Cádiz

IPD SHARING:
Plan to Share IPD: Yes
All data will be available in an open repository. RODIN is the Repository of Teaching and Research Objects of the University of Cádiz. It contributes to increased visibility of work developed, increases the impact and ensures the preservation of said production. All ethics aspects will be considered to ensure confidentiality of the data as detailed. The University of Cadiz has a new "hybrid cloud" infrastructure, made up of the University of Cadiz's own cloud, combined with others external providers. This service provides secure, efficient and reliable storage, which safeguards the necessary guarantees for autonomy, security and control over the data. Each researcher has an internal space of 500 GB, and an external cloud space of 250 GB. As for backup systems, the one offered by the UCA includes full copies of the space 3 times a week, while external providers have their own backup system, which allows restoring any accidentally deleted information up to 20 days after the incident.
Supporting Information: Study Protocol, SAP
URL: https://rodin.uca.es/handle/10498/6086

REFERENCES:
- [Background] Lowry KA, Vallejo AN, Studenski SA. Successful aging as a continuum of functional independence: lessons from physical disability models of aging. Aging Dis. 2012 Feb;3(1):5-15. Epub 2011 Aug 15. PMID 22500268
- [Background] Garcia-Garcia FJ, Larrion Zugasti JL, Rodriguez Manas L. [Frailty: a phenotype under review]. Gac Sanit. 2011 Dec;25 Suppl 2:51-8. doi: 10.1016/j.gaceta.2011.08.001. Epub 2011 Oct 26. Spanish. PMID 22033007
- [Background] Tavassoli N, Piau A, Berbon C, De Kerimel J, Lafont C, De Souto Barreto P, Guyonnet S, Takeda C, Carrie I, Angioni D, Paris F, Mathieu C, Ousset PJ, Balardy L, Voisin T, Sourdet S, Delrieu J, Bezombes V, Pons-Pretre V, Andrieu S, Nourhashemi F, Rolland Y, Soto ME, Beard J, Sumi Y, Araujo Carvalho I, Vellas B. Framework Implementation of the INSPIRE ICOPE-CARE Program in Collaboration with the World Health Organization (WHO) in the Occitania Region. J Frailty Aging. 2021;10(2):103-109. doi: 10.14283/jfa.2020.26. PMID 33575698
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838
- [Background] Warming L, Hassager C, Christiansen C. Changes in bone mineral density with age in men and women: a longitudinal study. Osteoporos Int. 2002;13(2):105-12. doi: 10.1007/s001980200001. PMID 11905520
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Berryman JW. Exercise is medicine: a historical perspective. Curr Sports Med Rep. 2010 Jul-Aug;9(4):195-201. doi: 10.1249/JSR.0b013e3181e7d86d. PMID 20622536
- [Background] Cadore EL, Izquierdo M. Exercise interventions in polypathological aging patients that coexist with diabetes mellitus: improving functional status and quality of life. Age (Dordr). 2015 Jun;37(3):64. doi: 10.1007/s11357-015-9800-2. Epub 2015 Jun 9. PMID 26054595
- [Background] Izquierdo M, Rodriguez-Manas L, Casas-Herrero A, Martinez-Velilla N, Cadore EL, Sinclair AJ. Is It Ethical Not to Precribe Physical Activity for the Elderly Frail? J Am Med Dir Assoc. 2016 Sep 1;17(9):779-81. doi: 10.1016/j.jamda.2016.06.015. Epub 2016 Jul 28. No abstract available. PMID 27477615
- [Background] Ahtiainen JP, Walker S, Peltonen H, Holviala J, Sillanpaa E, Karavirta L, Sallinen J, Mikkola J, Valkeinen H, Mero A, Hulmi JJ, Hakkinen K. Heterogeneity in resistance training-induced muscle strength and mass responses in men and women of different ages. Age (Dordr). 2016 Feb;38(1):10. doi: 10.1007/s11357-015-9870-1. Epub 2016 Jan 15. PMID 26767377
- [Background] Bonafiglia JT, Rotundo MP, Whittall JP, Scribbans TD, Graham RB, Gurd BJ. Inter-Individual Variability in the Adaptive Responses to Endurance and Sprint Interval Training: A Randomized Crossover Study. PLoS One. 2016 Dec 9;11(12):e0167790. doi: 10.1371/journal.pone.0167790. eCollection 2016. PMID 27936084
- [Background] Pickering, C. & Kiely, J. Understanding Personalized Training Responses: Can Genetic Assessment Help? Open Sports Sci. 2017; J 10, 191-213.
- [Background] Sarzynski MA, Ghosh S, Bouchard C. Genomic and transcriptomic predictors of response levels to endurance exercise training. J Physiol. 2017 May 1;595(9):2931-2939. doi: 10.1113/JP272559. Epub 2016 Jul 3. PMID 27234805
- [Background] Delmonico MJ, Kostek MC, Doldo NA, Hand BD, Walsh S, Conway JM, Carignan CR, Roth SM, Hurley BF. Alpha-actinin-3 (ACTN3) R577X polymorphism influences knee extensor peak power response to strength training in older men and women. J Gerontol A Biol Sci Med Sci. 2007 Feb;62(2):206-12. doi: 10.1093/gerona/62.2.206. PMID 17339648
- [Background] Charbonneau DE, Hanson ED, Ludlow AT, Delmonico MJ, Hurley BF, Roth SM. ACE genotype and the muscle hypertrophic and strength responses to strength training. Med Sci Sports Exerc. 2008 Apr;40(4):677-83. doi: 10.1249/MSS.0b013e318161eab9. PMID 18317377
- [Background] Espinosa-Salinas I, de la Iglesia R, Colmenarejo G, Molina S, Reglero G, Martinez JA, Loria-Kohen V, Ramirez de Molina A. GCKR rs780094 Polymorphism as A Genetic Variant Involved in Physical Exercise. Genes (Basel). 2019 Jul 28;10(8):570. doi: 10.3390/genes10080570. PMID 31357711
- [Background] Pickering C, Kiely J. ACTN3: More than Just a Gene for Speed. Front Physiol. 2017 Dec 18;8:1080. doi: 10.3389/fphys.2017.01080. eCollection 2017. PMID 29326606
- [Background] Pickering C, Kiely J. ACTN3, Morbidity, and Healthy Aging. Front Genet. 2018 Jan 24;9:15. doi: 10.3389/fgene.2018.00015. eCollection 2018. PMID 29416549
- [Background] Alibegovic AC, Sonne MP, Hojbjerre L, Bork-Jensen J, Jacobsen S, Nilsson E, Faerch K, Hiscock N, Mortensen B, Friedrichsen M, Stallknecht B, Dela F, Vaag A. Insulin resistance induced by physical inactivity is associated with multiple transcriptional changes in skeletal muscle in young men. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E752-63. doi: 10.1152/ajpendo.00590.2009. Epub 2010 Aug 24. PMID 20739510
- [Background] Tseng SH, Lee WJ, Peng LN, Lin MH, Chen LK. Associations between hemoglobin levels and sarcopenia and its components: Results from the I-Lan longitudinal study. Exp Gerontol. 2021 Jul 15;150:111379. doi: 10.1016/j.exger.2021.111379. Epub 2021 Apr 27. PMID 33930506
- [Background] Semba RD, Gonzalez-Freire M, Tanaka T, Biancotto A, Zhang P, Shardell M, Moaddel R; CHI Consortium; Ferrucci L. Elevated Plasma Growth and Differentiation Factor 15 Is Associated With Slower Gait Speed and Lower Physical Performance in Healthy Community-Dwelling Adults. J Gerontol A Biol Sci Med Sci. 2020 Jan 1;75(1):175-180. doi: 10.1093/gerona/glz071. PMID 30874790
- [Background] Kim M, Walston JD, Won CW. Associations Between Elevated Growth Differentiation Factor-15 and Sarcopenia Among Community-dwelling Older Adults. J Gerontol A Biol Sci Med Sci. 2022 Apr 1;77(4):770-780. doi: 10.1093/gerona/glab201. PMID 34255062
- [Background] Picca A, Guerra F, Calvani R, Marini F, Biancolillo A, Landi G, Beli R, Landi F, Bernabei R, Bentivoglio AR, Monaco MRL, Bucci C, Marzetti E. Mitochondrial Signatures in Circulating Extracellular Vesicles of Older Adults with Parkinson's Disease: Results from the EXosomes in PArkiNson's Disease (EXPAND) Study. J Clin Med. 2020 Feb 12;9(2):504. doi: 10.3390/jcm9020504. PMID 32059608
- [Background] McCarthy JJ. The MyomiR network in skeletal muscle plasticity. Exerc Sport Sci Rev. 2011 Jul;39(3):150-4. doi: 10.1097/JES.0b013e31821c01e1. PMID 21467943
- [Background] Liu HC, Han DS, Hsu CC, Wang JS. Circulating MicroRNA-486 and MicroRNA-146a serve as potential biomarkers of sarcopenia in the older adults. BMC Geriatr. 2021 Jan 30;21(1):86. doi: 10.1186/s12877-021-02040-0. PMID 33516190
- [Background] Cannataro R, Carbone L, Petro JL, Cione E, Vargas S, Angulo H, Forero DA, Odriozola-Martinez A, Kreider RB, Bonilla DA. Sarcopenia: Etiology, Nutritional Approaches, and miRNAs. Int J Mol Sci. 2021 Sep 8;22(18):9724. doi: 10.3390/ijms22189724. PMID 34575884
- [Background] Chang KV, Chen YC, Wu WT, Shen HJ, Huang KC, Chu HP, Han DS. Expression of Telomeric Repeat-Containing RNA Decreases in Sarcopenia and Increases after Exercise and Nutrition Intervention. Nutrients. 2020 Dec 8;12(12):3766. doi: 10.3390/nu12123766. PMID 33302352
- [Background] Galan-Mercant A, Baron-Lopez FJ, Labajos-Manzanares MT, Cuesta-Vargas AI. Reliability and criterion-related validity with a smartphone used in timed-up-and-go test. Biomed Eng Online. 2014 Dec 2;13:156. doi: 10.1186/1475-925X-13-156. PMID 25440533
- [Background] Cuesta-Vargas AI, Galan-Mercant A, Williams JM. The use of inertial sensors system for human motion analysis. Phys Ther Rev. 2010 Dec;15(6):462-473. doi: 10.1179/1743288X11Y.0000000006. PMID 23565045
- [Background] McGinley JL, Baker R, Wolfe R, Morris ME. The reliability of three-dimensional kinematic gait measurements: a systematic review. Gait Posture. 2009 Apr;29(3):360-9. doi: 10.1016/j.gaitpost.2008.09.003. Epub 2008 Nov 13. PMID 19013070
- [Background] Nawaratne R, Alahakoon D, De Silva D, O'Halloran PD, Montoye AH, Staley K, Nicholson M, Kingsley MI. Deep Learning to Predict Energy Expenditure and Activity Intensity in Free Living Conditions using Wrist-specific Accelerometry. J Sports Sci. 2021 Mar;39(6):683-690. doi: 10.1080/02640414.2020.1841394. Epub 2020 Oct 30. PMID 33121379
- [Background] Rockwood K, Abeysundera MJ, Mitnitski A. How should we grade frailty in nursing home patients? J Am Med Dir Assoc. 2007 Nov;8(9):595-603. doi: 10.1016/j.jamda.2007.07.012. Epub 2007 Oct 22. PMID 17998116
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Gruenewald TL, Seeman TE, Karlamangla AS, Sarkisian CA. Allostatic load and frailty in older adults. J Am Geriatr Soc. 2009 Sep;57(9):1525-31. doi: 10.1111/j.1532-5415.2009.02389.x. Epub 2009 Jul 21. PMID 19682116
- [Background] Losa-Reyna J, Baltasar-Fernandez I, Alcazar J, Navarro-Cruz R, Garcia-Garcia FJ, Alegre LM, Alfaro-Acha A. Effect of a short multicomponent exercise intervention focused on muscle power in frail and pre frail elderly: A pilot trial. Exp Gerontol. 2019 Jan;115:114-121. doi: 10.1016/j.exger.2018.11.022. Epub 2018 Dec 4. PMID 30528641
- [Background] Alcazar J, Losa-Reyna J, Rodriguez-Lopez C, Alfaro-Acha A, Rodriguez-Manas L, Ara I, Garcia-Garcia FJ, Alegre LM. The sit-to-stand muscle power test: An easy, inexpensive and portable procedure to assess muscle power in older people. Exp Gerontol. 2018 Oct 2;112:38-43. doi: 10.1016/j.exger.2018.08.006. Epub 2018 Sep 1. PMID 30179662
- [Background] Rodriguez-Lopez C, Alcazar J, Losa-Reyna J, Martin-Espinosa NM, Baltasar-Fernandez I, Ara I, Csapo R, Alegre LM. Effects of Power-Oriented Resistance Training With Heavy vs. Light Loads on Muscle-Tendon Function in Older Adults: A Study Protocol for a Randomized Controlled Trial. Front Physiol. 2021 Feb 18;12:635094. doi: 10.3389/fphys.2021.635094. eCollection 2021. PMID 33679447
- [Background] Losa-Reyna J, Alcazar J, Rodriguez-Gomez I, Alfaro-Acha A, Alegre LM, Rodriguez-Manas L, Ara I, Garcia-Garcia FJ. Low relative mechanical power in older adults: An operational definition and algorithm for its application in the clinical setting. Exp Gerontol. 2020 Dec;142:111141. doi: 10.1016/j.exger.2020.111141. Epub 2020 Oct 27. PMID 33127413
- [Background] Mateos-Angulo A, Galan-Mercant A, Cuesta-Vargas AI. Muscle thickness contribution to sit-to-stand ability in institutionalized older adults. Aging Clin Exp Res. 2020 Aug;32(8):1477-1483. doi: 10.1007/s40520-019-01328-x. Epub 2019 Aug 28. PMID 31463929
- [Derived] Mihaiescu-Ion V, Ortega-Gomez S, Dominguez-Navarro A, Ayala-Martinez C, Llerena-Guerrero R, Perez-Cabezas V, Gonzalez-Medina G, Losa-Reyna J, Galan-Mercant A. Viability of an educational program for lifestyle changes and an algorithm for the derivation of exercise programs in older people at risk of dependency at primary care: PRICA-POWFRAIL study protocol. BMC Geriatr. 2026 Feb 10. doi: 10.1186/s12877-025-06902-9. Online ahead of print. PMID 41663978